CLINICAL TRIAL: NCT00443547
Title: Prospective Multi-Center Clinical Study of Patients With Degenerative Disc Disease Treated With Anterior Cervical Decompression and Fusion Using the Vectra-T Translational Cervical Plate.
Brief Title: Outcome Study of Patients Treated With Translational Cervical Plate Used to Treat Degenerative Disc Disease
Status: Completed | Type: Observational
Sponsor: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VECTR 1492
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-06

CONDITIONS: Degenerative Disc Disease
Keywords: Prospective; Degenerative Disc Disease; Cervical; Translational Plate
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1-level: Patients needing a single level cervical fusion with Vectra-T
  Interventions: Device: Vectra-T
- 2-level: Patients needing cervical fusion at two consecutive levels with Vectra-T
  Interventions: Device: Vectra-T
- 3-level: Patients needing cervical fusion at three consecutive levels with Vectra-T
  Interventions: Device: Vectra-T
- 4-level: Patients needing cervical fusion at four consecutive levels with Vectra-T
  Interventions: Device: Vectra-T

INTERVENTIONS:
Device: Vectra-T — Patient will receive the Vectra-T plate (Sized 1 to 4 levels)
  Other Names: Vectra-T Translational Plating System

SUMMARY:
The purpose of this study is to measure the benefits of anterior (from the front) cervical (neck) surgery for degenerative disc disease. The research part of this study is the answering of questionnaires by the patient concerning their quality of life, prior to, and after surgery.

DETAILED DESCRIPTION:
This is a prospective, multi-center, four-arm study designed to evaluate the clinical and radiographic outcomes in patients diagnosed with cervical degenerative disc disease (DDD) and treated using the Vectra-T Cervical Plate and the Advanced ACF or CorticoCancellous Allograft Spacer made by Synthes Spine Company (Paoli, PA). This is not an investigational study (IDE) and no investigational or experimental devices or procedures are included in this study.

ELIGIBILITY:
Inclusion Criteria:

* One to four levels (consecutive) cervical degenerative disc disease between C2 and C7, defined as at least one of the following:

  * disc herniation
  * axial neck pain (with or without radiculopathy or myelopathy) caused by spondylosis
  * functional deficit
  * neurological deficit which significantly limits patient's normal living
* One to four cervical levels to be plated
* Patient is skeletally mature and at least 18 years of age
* Patient signs consent form
* Patient is available for long term (24 month) follow-up
* Etiology must be confirmed by MRI or CT

Exclusion Criteria:

* Spondylolisthesis greater than grade 1 at either level(s) to be instrumented
* Indications for complete corpectomy of any involved levels
* Posterior instrumentation is necessary at same levels
* More than one previous failed anterior fusion attempt at the involved level(s)
* Has had more than one previous open, posterior, spine surgical procedures at the involved level(s) or pre-op instability on Flexion/Extension radiographs.
* Pregnant or interested in becoming pregnant during the study follow-up period
* Has a known sensitivity to device materials
* Mentally incompetent or prisoner
* Currently a participant in a study related to the treatment of cervical spinal disorders
* Pre-op instability>3mm on flexion/extension X-rays

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgeon's personal patient contacts
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2006-03-01 (Actual); Primary Completion 2011-04-01 (Actual); Study Completion 2011-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Kovalsky, M.D., Principal Investigator
Locations (13):
- United States (13):
  - Roderick Sanden, MD, Carmichael, California
  - Yu-Po Lee, MD, La Jolla, California
  - Ardavan Aslie, MD, Marysville, California
  - Barry Chehrazi, MD, Roseville, California
  - Don Kovalsky, MD, Mount Vernon, Illinois
  - Mark Crawford, MD, Fort Wayne, Indiana
  - Faheem Sandhu, MD, Clinton, Maryland
  - Chris Urban, MD, Glen Burnie, Maryland
  - John Moriarity, MD, Flowood, Mississippi
  - Jamal Taha, MD, Kettering, Ohio
  - Abhay Varma, MD, Charleston, South Carolina
  - Daniel Nehls, MD, Tacoma, Washington
  - Dennis Maiman, MD, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-level: Patients needing a single level cervical fusion with Vectra-T Vectra-T: Patient will receive the Vectra-T plate (Sized 1 to 4 levels)
- 2-level: Patients needing cervical fusion at two consecutive levels with Vectra-T Vectra-T: Patient will receive the Vectra-T plate (Sized 1 to 4 levels)
- 3-level: Patients needing cervical fusion at three consecutive levels with Vectra-T Vectra-T: Patient will receive the Vectra-T plate (Sized 1 to 4 levels)
- 4-level: Patients needing cervical fusion at four consecutive levels with Vectra-T Vectra-T: Patient will receive the Vectra-T plate (Sized 1 to 4 levels)
Period: Overall Study
Arm/Group | 1-level | 2-level | 3-level | 4-level
Started | 89 (Enrolled and Treated Per Protocol) | 88 (Enrolled and Treated Per Protocol) | 48 (Enrolled and Treated Per Protocol) | 6 (Enrolled and Treated Per Protocol)
Evaluated at 12 Months | 58 | 55 | 37 | 5
Completed | 44 | 46 | 27 | 4
Not Completed | 45 | 42 | 21 | 2

BASELINE CHARACTERISTICS:
Population: Subjects Enrolled and Treated Per Protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-level | 2-level | 3-level | 4-level | Total
Number analyzed (Participants) | 89 | 88 | 48 | 6 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age and Gender was not available for two (2) subjects. These subjects were treated at 1 and 2 Levels respectively.
  years
    number analyzed (Participants) | 88 | 87 | 48 | 6 | 229
    (all) | 46.8 (10.58) | 50.3 (9.6) | 55.8 (11.4) | 56.4 (12.1) | 50.8 (12.1)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Gender was not reported for 2 Subjects; 1 at Level 1 and 1 at Level 2. Number analyzed will differ from other reported populations
  Participants
    number analyzed (Participants) | 88 | 87 | 48 | 6 | 229
    Female | 43 | 49 | 29 | 5 | 126
    Male | 45 | 38 | 19 | 1 | 103
Region of Enrollment [Count of Participants; unit: Participants]
  United States: United States | 89 | 88 | 48 | 6 | 231
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI unit of measure is kg/m^2
  kg/m^2 | 29.3 (6.0) | 29.2 (6.0) | 28.8 (5.5) | 35.9 (13.9) | 29.3 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Fusion
Description: Percentage of subjects who were successfully fused per an independent radiographic assessment at all index levels
Time Frame: 24 Months
Population: Number of subjects present for the 24 month visit
Measure: Number; unit: percentage of subjects
Arm/Group | 1-level | 2-level | 3-level | 4-level
Number analyzed (Participants) | 44 | 46 | 27 | 4
percentage of subjects | 66 | 46 | 37 | 75

2. Primary Outcome: Radiographic Fusion
Description: Percentage of subjects who were successfully fused per an independent radiographic assessment at all index levels
Time Frame: 12 Months
Population: Number of subjects present for the 12 month visit
Measure: Number; unit: percentage of subjects
Arm/Group | 1-level | 2-level | 3-level | 4-level
Number analyzed (Participants) | 58 | 55 | 37 | 5
percentage of subjects | 48 | 25 | 27 | 20

3. Secondary Outcome: Neck Disability Index (NDI) is a Widely Used Instrument for Assessing Self-reported Disability in Patients With Neck Pain. Scoring is Reported on a 0-100 Point Scale, 0 Being the Best Possible Score and 100 Being the Worst Possible Score
Description: Average NDI score at 24 months - score range is 0 to 100, with 0 being the best and 100 being the worst
Time Frame: 24 Months
Population: The Total Population enrolled and treated includes 89 (1-Level), 88 (2-Level), 48 (3-Level), and 6 (4-Level). With each outcome measure, the actual Overall Number of Participants Analyzed will vary based on the actual number of participants who completed the specific assessment at the specific timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1-level | 2-level | 3-level | 4-level
Number analyzed (Participants) | 42 | 47 | 27 | 5
units on a scale | 27 (22) | 29 (21) | 24 (22) | 17 (16)

ADVERSE EVENTS:
Time Frame: From enrollment through 24 months
Arm/Group | 1-level | 2-level | 3-level | 4-level
Serious Adverse Events (participants affected / at risk) | 3/89 | 1/88 | 0/48 | 0/6
Other Adverse Events (participants affected / at risk) | 8/89 | 13/88 | 5/48 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-level (N=89) | 2-level (N=88) | 3-level (N=48) | 4-level (N=6)
Non-Union (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-level (N=89) | 2-level (N=88) | 3-level (N=48) | 4-level (N=6)
Hematoma / Seroma (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neurological Deficit (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Nervous system disorders) | 4 (5) | 4 (4) | 2 (2) | 0 (0)
Non-Union (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Numbness or Tingling (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Other (General disorders) | 4 (4) | 3 (3) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less